CLINICAL TRIAL: NCT06196281
Title: Effects of Multi Station Proprioceptive Training in Soccer Players With Hamstrings Strain
Brief Title: Multi Station Training in Soccer Players Hamstrings Strain
Acronym: EMPTSPHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0448
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Sports Physical Therapy
Keywords: multistation proprioceptive training; soccer players; hamstrings strain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wooble board proprioceptive training (Experimental): The group A will perform the wobble board proprioceptive training program lasting for four weeks. Both the training programs consisted of one-leg and double-leg static and dynamic balance drills
  Interventions: Other: wooble board proprioceptive training; Other: multi-station proprioceptive training
- multi-station proprioceptive training (Experimental): The group B will perform the multi-station proprioceptive training program lasting for four weeks. Both the training programs consisted of one-leg and double-leg static and dynamic balance drills basic exercise single length stance walk, Jumper exercise, resistance exercise
  Interventions: Other: wooble board proprioceptive training; Other: multi-station proprioceptive training

INTERVENTIONS:
Other: wooble board proprioceptive training — this includes wooble board proprioceptive training twice a day for four weeks
  Other Names: wooble board training
Other: multi-station proprioceptive training — this includes multi-station proprioceptive training twice a day for four weeks
  Other Names: multi-station training

SUMMARY:
The study is a randomized controlled trial. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Group A will be the wobble board proprioceptive training program lasting for four weeks, while Group B will be administered the multi-station proprioceptive training program lasting for four weeks.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of Multi-station Proprioceptive training on hamstring strains in Soccer Players. The study is a randomized controlled trial. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Group A will be the wobble board proprioceptive training program lasting for four weeks, while Group B will be administered the multi-station proprioceptive training program lasting for four weeks. Outcome measures will be assessed by using NPRS, Sit And Reach Test. Lower Extremity Functional Scale. Proximal Hamstring Injury Questionnaire. Balance Training Tool. The collected data will be analyzed in statistical Package for the social Sciences (SPSS) 25.0 .Parametric ∕non|-parametric tests will be applied after test normality of data

ELIGIBILITY:
Inclusion Criteria:

* Male football players (trained - not trained) between 14 and 30 years of age, Players with a history of hamstring strain had reduced SLH scores, Players with a history of right knee injury also had reduced SLHB scores on the injured side

Exclusion Criteria:

* Children and older adults, Upper body proprioceptive training, Presence of pain in any part of upper limb,lower limb, trunk or body which can interfere in training session

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | pre and 4 weeks post intervention
  pain will be measured by Numeric Pain Rating Scale (NPRS)
Hamstrings and low back flexibility | pre and post 4 weeks intervention
  Sit and Reach test will be used to measure hamstrings and low back flexibility
Activities of daily living | pre and post 4 weeks intervention
  lower extremity functional scale is used to measure ability to perform activities of daily living
Single limb stance excursion distances | pre and post 4 weeks intervention
  Y balance test will be used to measure single limb stance excursion distances

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abbas, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abian-Vicen J, Alegre LM, Fernandez-Rodriguez JM, Aguado X. Prophylactic ankle taping: elastic versus inelastic taping. Foot Ankle Int. 2009 Mar;30(3):218-25. doi: 10.3113/FAI.2009.0218. PMID 19321098
- [Background] Akbari A, Sarmadi A, Zafardanesh P. The effect of ankle taping and balance exercises on postural stability indices in healthy women. J Phys Ther Sci. 2014 May;26(5):763-9. doi: 10.1589/jpts.26.763. Epub 2014 May 29. PMID 24926148
- [Background] Leiva JJA. Propuesta de incorporación de tareas preventivas basadas en métodos propioceptivos en fútbol. Retos: nuevas tendencias en educación física, deporte y recreación. 2014(26):163-7
- [Background] Márquez Arabia JJ, Ramón Suárez G, Quiceno Noguera C. Lesiones en futbolistas de un equipo sudamericano durante 1 año de seguimiento. Revista Cubana de Ortopedia y Traumatología. 2016;30(1):65-75.
- [Background] Villaquirán AF, Dorado EP, Vernaza P. Caracterización de la lesión deportiva en atletas caucanos con proyección a Juegos Deportivos Nacionales. Universidad y salud. 2016;18(3):541-9.
- [Background] Schiftan GS, Ross LA, Hahne AJ. The effectiveness of proprioceptive training in preventing ankle sprains in sporting populations: a systematic review and meta-analysis. J Sci Med Sport. 2015 May;18(3):238-44. doi: 10.1016/j.jsams.2014.04.005. Epub 2014 Apr 26. PMID 24831756
- [Background] Gaurav S, Pooja A, Shishir N, Tanvi A. Comparative analysis of effectiveness of conventional proprioceptive training and multistation proprioceptive training on vertical jump performance in Indian basketball players. Journal of Exercise Science and Physiotherapy. 2013;9(2):97-104.
- [Background] Cerulli G, Benoit DL, Caraffa A, Ponteggia F. Proprioceptive training and prevention of anterior cruciate ligament injuries in soccer. J Orthop Sports Phys Ther. 2001 Nov;31(11):655-60; discussion 661. doi: 10.2519/jospt.2001.31.11.655. PMID 11720298
- [Background] Kennedy JC, Alexander IJ, Hayes KC. Nerve supply of the human knee and its functional importance. Am J Sports Med. 1982 Nov-Dec;10(6):329-35. doi: 10.1177/036354658201000601. PMID 6897495
- [Background] Ogard WK. Proprioception in sports medicine and athletic conditioning. Strength & Conditioning Journal. 2011;33(3):111-8.
- [Background] Lizardo FB, Ronzani GM, Sousa LR, Silva DCdO, Santos LAd, Lopes PR, et al. Proprioceptive exercise with bosu maximizes electromyographic activity of the ankle muscles. Biosci j(Online). 2017:754-62.
- [Background] Lephart SM, Pincivero DM, Giraldo JL, Fu FH. The role of proprioception in the management and rehabilitation of athletic injuries. Am J Sports Med. 1997 Jan-Feb;25(1):130-7. doi: 10.1177/036354659702500126. PMID 9006708
- [Background] Valentin S, Linton L, Sculthorpe NF. Effect of supervision and athlete age and sex on exercise-based injury prevention programme effectiveness in sport: A meta-analysis of 44 studies. Res Sports Med. 2024 Sep-Oct;32(5):705-724. doi: 10.1080/15438627.2023.2220059. Epub 2023 Jun 7. PMID 37283040
- [Background] Brunn H, Arnold G, Körner W, Rippen G, Steinhäuser KG, Valentin I. PFAS: forever chemicals-persistent, bioaccumulative and mobile. Reviewing the status and the need for their phase out and remediation of contaminated sites. Environmental Sciences Europe. 2023;35(1):1-50.
- [Background] Akerlund I, Walden M, Sonesson S, Hagglund M. Forty-five per cent lower acute injury incidence but no effect on overuse injury prevalence in youth floorball players (aged 12-17 years) who used an injury prevention exercise programme: two-armed parallel-group cluster randomised controlled trial. Br J Sports Med. 2020 Sep;54(17):1028-1035. doi: 10.1136/bjsports-2019-101295. Epub 2020 Jan 28. PMID 31992545
- [Background] Fischer F, Fink C, Herbst E, Hoser C, Hepperger C, Blank C, Gfoller P. Higher hamstring-to-quadriceps isokinetic strength ratio during the first post-operative months in patients with quadriceps tendon compared to hamstring tendon graft following ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2018 Feb;26(2):418-425. doi: 10.1007/s00167-017-4522-x. Epub 2017 Mar 21. PMID 28324151
- [Background] van Doormaal MC, van der Horst N, Backx FJ, Smits DW, Huisstede BM. No Relationship Between Hamstring Flexibility and Hamstring Injuries in Male Amateur Soccer Players: A Prospective Study. Am J Sports Med. 2017 Jan;45(1):121-126. doi: 10.1177/0363546516664162. Epub 2016 Oct 1. PMID 27582278
- [Background] Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Reprint--preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. Phys Ther. 2009 Sep;89(9):873-80. No abstract available. PMID 19723669
- [Background] Breivik EK, Bjornsson GA, Skovlund E. A comparison of pain rating scales by sampling from clinical trial data. Clin J Pain. 2000 Mar;16(1):22-8. doi: 10.1097/00002508-200003000-00005. PMID 10741815
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543